CLINICAL TRIAL: NCT03413319
Title: Extension Study of ABBV-8E12 in Patients With Progressive Supranuclear Palsy (PSP) Who Completed Study C2N-8E12-WW-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-948
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Progressive Supranuclear Palsy (PSP)
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — tilavonemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-8E12 (Experimental): ABBV-8E12 administered by intravenous (IV) infusion.
  Interventions: Drug: ABBV-8E12

INTERVENTIONS:
Drug: ABBV-8E12 — Solution for infusion
  Other Names: Tilavonemab

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of ABBV-8E12 in subjects with progressive supranuclear palsy (PSP).

ELIGIBILITY:
Inclusion Criteria:

* Subject completed Study C2N-8E12-WW-104 (NCT02494024)
* Subject was not eligible to enroll in Study M15-562 (NCT02985879)

Exclusion Criteria:

* Subject weighs less than 35 kg at screening
* Subject has any contraindication or inability to tolerate brain MRI
* Subject has any significant change in his/her medical condition that could interfere with the subject's participation in the study, could place the subject at increased risk, or could confound interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From first dose of study drug to 20 weeks after last dose of study drug (up to 2 years, 5 months)
  Adverse events and serious adverse events will be monitored throughout the dosing period and for approximately 20 weeks after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (2):
- United States (2):
  - University of California, San /ID# 170113, La Jolla, California
  - Texas Health Physicians Group /ID# 170112, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No